CLINICAL TRIAL: NCT00916877
Title: Prophylactic Cranial Irradiation in Patients With HER-2-Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alberta Health services (Other)
Responsible Party: Drs Abdulkarim, Gabos and Mackey, Cross Cancer Institute
Organization: AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Inhouse
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: Prophylactic Cranial Irradiation; Her-2-positive met breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Prophylactic Cranial Irradiation — Prophylactic Cranial Irradiation

SUMMARY:
Though brain metastases are a risk in all patients with breast cancer, those with HER-2 overexpression are at significantly greater risk. One series estimated a 30% incidence of brain metastases in this population, while another study found an incidence of approximately 40%. Traditional systemic therapies do not cross the blood brain barrier to any significant degree or at all, but radiation treatment can be effective in the treatment of intracranial metastases.

DETAILED DESCRIPTION:
The rationale for PCI is that the brain is a sanctuary site where cancer cells can remain inaccessible to chemotheraphy and agents such as trastuzumab due to the blood brain barrier, which prevents potentially harmful chemicals such as chemotherapy agents and antibodies such as trastuzumab from reaching the brain. Decreasing the incidence of brain metastasis with acceptable effects on neurocognitive function would be a significant improvement in the care of patients with MBC.

ELIGIBILITY:
Inclusion Criteria:

* Female with HER2-positive disease
* 18 years of age or older
* ECOG greater or equal to 2
* Life expectancy greater or equal to 6 months
* Able to complete self administered quality of life evaluations and neurocognitive testing
* Willing and able to comply with study instructions and commit to all clinic visits for the duration of the study
* Women of child-bearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at the baseline visit and must use highly effective birth control during study
* Signed informed consent form

Exclusion Criteria:

* Current malignancy in the brain, as determined by screening MRI/CT done no more then 6 weeks prior to study treatment with PCI
* Chemo or radiation planned during the period when patients will receive study treatment with PCI
* Prior radiotherapy of the brain
* Prior stroke or brain hemorrhage in the 6 months prior to screening
* History of neurological/psychiatric disorders, including psychotic disorders or demential, or any other reason, which may affect neurocognitive assessment
* Inadequate renal function
* Other known previous or concomitant serious illness or medical condition that may interfere with participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of PCI, specifically with respect to neurocognitive function in patients with HER-2-positive metastatic breast cancer. | approximately 2 to 3 years from study start

SECONDARY OUTCOMES:
To assess the impact of PCI on measures of survival, specifically brain metastases-free survival, overall progression free survival and overall survival | approximately 4 years from study start

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada